CLINICAL TRIAL: NCT06765213
Title: Evaluation of Human Breast Milk and Its Role in Early Food Allergen Sensitization in Infants
Brief Title: Human Breast Milk's Role in Food Allergy Development
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Texas Allergy, Asthma, and Immunology Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22-0307
Record Dates: First submitted 2024-12-23; First posted 2025-01-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Food Allergy in Infants; Food Allergen Sensitisation; Breast Feeding, Exclusive; Breastmilk Collection
Keywords: food allergy; breastmilk allergen testing; food allergen sensitization; cow milk allergy; egg allergy; wheat allergy
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression; Food Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity; Wheat Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Breastmilk positive/Infant sensitized: This group is for infants whose mother's breastmilk is found to be positive for allergens to either cow milk, egg, and/or wheat and who are found to be sensitized to one or more of these allergens.
  Interventions: Diagnostic Test: Open Ended Oral Food Challenge
- Breastmilk positive/Infant not sensitized: This group is for infants whose mother's breastmilk is found to be positive for allergens to either cow milk, egg, and/or wheat and who are found to be not sensitized to the three allergens.
  Interventions: Other: Early Introduction
- Breastmilk negative/Infant sensitized: This group is for infants whose mother's breastmilk is found to be negative for allergens to either cow milk, egg, and/or wheat and who are found to be sensitized to one or more of these allergens.
  Interventions: Diagnostic Test: Open Ended Oral Food Challenge
- Breastmilk negative/Infant not sensitized: This group is for infants whose mother's breastmilk is found to be negative for allergens to either cow milk, egg, and/or wheat and who are found to be not sensitized to the three allergens.
  Interventions: Other: Early Introduction

INTERVENTIONS:
Diagnostic Test: Open Ended Oral Food Challenge — Allergens determined to be sensitized will be brought in for an oral challenge to that food.
  Groups: Breastmilk negative/Infant sensitized; Breastmilk positive/Infant sensitized
Other: Early Introduction — Infants that are not sensitized will have the food introduced to their diet at regular intervals.
  Groups: Breastmilk negative/Infant not sensitized; Breastmilk positive/Infant not sensitized

SUMMARY:
The goal of this prospective cohort pilot study is to learn about food allergens being passed on in breast milk to breast feeding infants.

The main question[s] it aims to answer are:

* Will major allergens for milk, egg, and peanut be passed on to infants in breast milk?
* Will the infants become sensitized to and develop an allergy to the food allergens found in breast milk?
* Will early introduction interventions prevent the development of these food allergies?

Participants will

* provide breast milk sample (s) for testing for food allergens
* Infants will be tested for sensitization via skin prick and blood testing
* Infants will be challenge with suspected foods to determine allergy and undergo early introduction procedures

DETAILED DESCRIPTION:
Recruitment of subjects will be open enrollment pregnant or post-partum women with a personal history of atopic disease such as allergic rhinitis/conjunctivitis, asthma, atopic dermatitis (eczema), and/or food allergy who are exclusively breastfeeding.

Mothers will provide a breastmilk sample(s) for testing of allergens to milk, egg, and wheat. Prior to the introduction of solid foods, infants will need to be tested for sensitization to milk, egg, and wheat via skin prick testing and blood allergy testing.

Infants that are negative for sensitization will undergo introduction of these foods per standard practice. Infants that are positive for sensitization will undergo an office food challenge for those foods that they are sensitized to. A positive food challenge is diagnostic for a food allergy and they will be managed according to standard practice. A negative food challenge means that they are not allergic, and they will undergo early introduction protocols and monitored to continued tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant or post-partum females who plan to exclusively breastfeed and their infants who have completed at least 37 weeks of gestation

   1. These are vulnerable populations
   2. Our study involves breastmilk analysis, which we need postpartum mothers to supply.
   3. (Parent) Testing will be done solely on breastmilk samples, with only potential dietary intervention done to the parent postpartum depending on the outcomes of the infant and breastmilk.
   4. (Infant) In order to determine if allergens in breastmilk play a role in food allergen sensitization, we need to test the infants prior to the introduction of solid foods.
2. Personal history of atopic disease such as allergic rhinitis/conjunctivitis, asthma, food allergies, and atopic dermatitis
3. Maternal diet must include hen's egg, cow's milk, and wheat products.

Exclusion Criteria:

1. No maternal history of atopic disease
2. Exclusive formula feeding
3. Maternal diet devoid of hen's egg, cow's milk, or wheat, for example, vegan diets and persons with gluten sensitivity.

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants at 4 months of age up to 24 months of age.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the detection of allergens in human breast milk | Baseline (4 months of age)
  A mass spectrometry will be used to detect the allergens. Mass spectrometry is a technique used in the University of Texas Medical Branch (UTMB) laboratory to detect allergens.
To assess breast milk's role in sensitization to allergens | Baseline (4 months of age)
  The infant will be skin prick tested for allergens to milk, eggs, and wheat at 4 months, which is the baseline.

SECONDARY OUTCOMES:
Number of non-sensitized participants | Baseline (4 months of age), 12 months of age, 24 months of age
  The infants that are non-sensitized will begin consuming milk, eggs, and wheat, and each well child check visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Sub Specialty Clinic at Bay Colony, League City, Texas, United States

IPD SHARING:
Plan to Share IPD: No